CLINICAL TRIAL: NCT04175834
Title: Comparing the Risk and Severity of Infusion-Related Reactions in Patients Premedicated With Cetirizine Versus Diphenhydramine Prior to Ocrelizumab Infusions
Brief Title: Comparing Risk and Severity of IRRs in Patients Premedicated With Cetirizine vs. Diphenhydramine Prior to Ocrelizumab
Acronym: PRECEPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML41308; PRECEPT (Other: Providence health & Services)
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis; Infusion Reaction
Keywords: cetirizine; diphenhydramine
MeSH Terms: conditions — Multiple Sclerosis | interventions — Diphenhydramine

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, pilot study to determine there is evidence that cetirizine is non-inferior to diphenhydramine in limiting the proportion and severity of infusion related reactions to ocrelizumab infusions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- diphenhydramine (Other): 25 mg diphenhydramine capsule, generic, sourced from Major Pharmaceuticals will be give orally 30-60 minutes prior to ocrelizumab infusion.
  Interventions: Drug: diphenhydramine
- cetirizine (Active Comparator): 10 mg cetirizine tablet, generic, sourced from Mylan Pharmaceuticals will be give orally 30-60 minutes prior to ocrelizumab infusion.
  Interventions: Drug: cetrizine

INTERVENTIONS:
Drug: cetrizine — prophylaxis
  Other Names: Active comparator
  Arms: cetirizine
Drug: diphenhydramine — prophylaxis
  Other Names: Other
  Arms: diphenhydramine

SUMMARY:
This 6-month randomized controlled pilot study will determine whether there is some evidence that cetirizine is better tolerated than diphenhydramine without an increase in Infusion-Related Reactions (IRRs) in subjects receiving ocrelizumab(OCR) for multiple sclerosis (MS).

DETAILED DESCRIPTION:
Ocrelizumab was approved by the US Food and Drug administration in March 2017 for the indication of Relapsing Remitting Multiple Sclerosis (RRMS) and Primary Progressive Multiple Sclerosis (PPMS). The landmark studies used to gain approval found ocrelizumab (OCR) to be well tolerated, but that at least one Infusion-Related Reaction (IRR) occurred in about one-third of patients. Because of this, neurologists typically prescribe prophylactic premedication with 100mg of methylprednisolone, 1 gram of acetaminophen, and 50 mg of IV diphenhydramine. However, many patients experience extreme sedation that interferes with their lifestyle considerably.

This 6-month randomized controlled pilot study will determine whether there is some evidence that cetirizine is better tolerated than diphenhydramine without an increase in IRRs. Fifty-two patients, 26 patients per arm, will be randomized in a 1:1 ratio to receive cetirizine or diphenhydramine as premedication prior to OCR infusions on day 0 (1st half dose of 300mg), day 14 (2nd half dose of 300mg) and week 24 (1st full dose of 600mg).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient with relapsing or progressive forms of Multiple Sclerosis (MS), age 18 to 70 inclusive at the time of consent.
2. Able to understand the purpose, responsibilities and risks of the study and provide signed informed consent.
3. Naïve to ocrelizumab (OCR) and will receive OCR as part of standard of care for MS treatment.
4. No evidence, in the opinion of the investigators of significant cognitive limitation or psychiatric disorder that would interfere with the conduct of the study.
5. Estimated Expanded Disability Status Scale (EDSS) of ≤ 6.5 at screening.
6. Female patients of childbearing potential must practice effective contraception and continue contraception during the study.

Exclusion Criteria:

1. Any mental condition of such that patient is unable to understand the nature, scope, and possible consequences of the study.
2. Evidence of active hepatitis B infection at screening.
3. Patients with untreated hepatitis C, or tuberculosis. Patients who have history of Progressive multifocal leukoencephalopathy (PML) or known to be Human Immunodeficiency Virus (HIV) positive, per standard care.
4. Any persistent or severe infection.
5. Pregnancy or lactation.
6. Significant, uncontrolled somatic disease or severe depression in the last year.
7. Current use of immunosuppressive medication, lymphocyte-depleting agents, or lymphocyte-trafficking blockers.
8. Patients with any significant comorbidity that in the opinion of the investigator, would interfere with participation in the study.
9. Any known allergy or inability to tolerate diphenhydramine or cetirizine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Smoot, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Neurological Specialties West, Portland, Oregon, United States

REFERENCES:
- [Background] National Cancer Institute. Common Terminology Criteria for Adverse Events (CTCAE). https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm. Accessed 02/13/19, 2019.
- [Background] Genentech Inc. Ocrevus: Highlights of Prescribing Information. 2018; https://www.gene.com/download/pdf/ocrevus_prescribing.pdf. Accessed 02/13/2019.
- [Background] Mylan Pharmaceuticals. cetirizine hydrochloride 10 mg tablet. https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=bd0dc7f6-5fb9-4381-bd81-b150b75a2c68. Accessed 9/3/2019, 2019.
- [Background] Major Pharmaceuticals. diphenhydramine hydrochloride 25mg capsule. https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=04e70311-6412-4a20-84e3-f6e26d5f19ab. Accessed 9/3/2019, 2019.
- [Background] US Food and Drug Administration. Non-Inferiority Clinical Trials to Establish Effectiveness: Guidance for Industry. 2016.
- [Result] Hauser SL, Bar-Or A, Comi G, Giovannoni G, Hartung HP, Hemmer B, Lublin F, Montalban X, Rammohan KW, Selmaj K, Traboulsee A, Wolinsky JS, Arnold DL, Klingelschmitt G, Masterman D, Fontoura P, Belachew S, Chin P, Mairon N, Garren H, Kappos L; OPERA I and OPERA II Clinical Investigators. Ocrelizumab versus Interferon Beta-1a in Relapsing Multiple Sclerosis. N Engl J Med. 2017 Jan 19;376(3):221-234. doi: 10.1056/NEJMoa1601277. Epub 2016 Dec 21. PMID 28002679
- [Result] Montalban X, Hauser SL, Kappos L, Arnold DL, Bar-Or A, Comi G, de Seze J, Giovannoni G, Hartung HP, Hemmer B, Lublin F, Rammohan KW, Selmaj K, Traboulsee A, Sauter A, Masterman D, Fontoura P, Belachew S, Garren H, Mairon N, Chin P, Wolinsky JS; ORATORIO Clinical Investigators. Ocrelizumab versus Placebo in Primary Progressive Multiple Sclerosis. N Engl J Med. 2017 Jan 19;376(3):209-220. doi: 10.1056/NEJMoa1606468. Epub 2016 Dec 21. PMID 28002688

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients with relapsing or progressive multiple sclerosis (MS), starting ocrelizumab (OCR)
Groups:
- Diphenhydramine: 25 mg diphenhydramine capsule, generic, sourced from Major Pharmaceuticals will be given orally 30-60 minutes prior to ocrelizumab infusion.
  antihistamine: prophylaxis
- Cetirizine: 10 mg cetirizine tablet, generic, sourced from Mylan Pharmaceuticals will be given orally 30-60 minutes prior to ocrelizumab infusion.
  antihistamine: prophylaxis
Period: Overall Study
Arm/Group | Diphenhydramine | Cetirizine
Started | 9 | 10
Completed | 8 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Diphenhydramine: 25 mg diphenhydramine capsule, generic, sourced from Major Pharmaceuticals will be give orally 30-60 minutes prior to ocrelizumab infusion.
  antihistamine: prophylaxis
- Cetirizine: 10 mg cetirizine tablet, generic, sourced from Mylan Pharmaceuticals will be give orally 30-60 minutes prior to ocrelizumab infusion.
  antihistamine: prophylaxis
- Total: Total of all reporting groups
Arm/Group | Diphenhydramine | Cetirizine | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (12.3) | 37.4 (9.40) | 36.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 8 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 10 | 19
Age at MS symptoms onset [Median (Inter-Quartile Range); unit: years] | 33.9 [30.0 to 36.5] | 33.7 [29.5 to 47.0] | 33.9 [19.4 to 56.4]
Age at MS diagnosis [Median (Inter-Quartile Range); unit: years] | 36.7 [30.1 to 45.3] | 34.5 [29.6 to 47.1] | 34.6 [19.8 to 63.1]
From MS symptoms onset to MS Diagnosis [Median (Inter-Quartile Range); unit: weeks] | 8.6 [5.4 to 209] | 7.4 [2.5 to 25.9] | 8.6 [0 to 465]
Age at OCR start [Median (Inter-Quartile Range); unit: years] | 46.3 [39.8 to 52.2] | 48.2 [38.0 to 54.0] | 47.5 [29.0 to 63.2]
Education [Count of Participants; unit: Participants]
  High School | 1 | 1 | 2
  Trade School | 1 | 0 | 1
  Associate's Degree | 4 | 1 | 5
  Bachelor's Degree | 3 | 5 | 8
  Graduate School | 0 | 3 | 3
Employment [Count of Participants; unit: Participants]
  Disabled | 1 | 1 | 2
  Full-time | 7 | 5 | 12
  Not working | 0 | 4 | 4
  Retired | 1 | 0 | 1
MS Type [Count of Participants; unit: Participants] — Participants are categorized as having Primary Progressive Multiple Sclerosis (PPMS), Relapsing-Remitting Multiple Sclerosis (RMS), or Secondary Progressive Multiple Sclerosis (SPMS) based on the review of their disease and medical history.
  Participants
    Primary Progressive Multiple Sclerosis (PPMS) | 1 | 0 | 1
    Relapsing-Remitting Multiple Sclerosis (RRMS) | 6 | 10 | 16
    Secondary Progressive Mutiple Sclerosis (SPMS) | 2 | 0 | 2
Reason start OCR [Count of Participants; unit: Participants]
  Breakthrough disease activity on previous treatment | 3 | 5 | 8
  Convenience | 2 | 0 | 2
  First-line therapy | 2 | 3 | 5
  Risk reduction from prior treatment | 2 | 1 | 3
  Side effects of prior treatment | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Infusion-related Reaction (IRR) on Day 0
Description: The proportion of patients having an infusion-related reaction (IRR), as defined by Common Terminology Criteria (CTCAE), version 4 during or after the first-half dose of the first infusion on day 0. IRRs are documented at the infusion clinic on the day of infusion and reported by the patient at the follow-up phone call the next business day after the infusion.
Time Frame: During or after the first-half dose of the first infusion on day 0
Measure: Number; unit: participnats
Arm/Group | Diphenhydramine | Cetirizine
Number analyzed (Participants) | 9 | 10
participnats | 5 | 6

2. Secondary Outcome: Proportion of Participants With Infusion-related Reaction (IRR) on Day 14
Description: The proportion of patients having an infusion-related reaction as defined by Common Terminology Criteria (CTCAE), version 4 during or after receiving the second half dose infusion on day 14
Time Frame: during or after receiving the second half dose infusion on day 14.
Measure: Number; unit: participants
Arm/Group | Diphenhydramine | Cetirizine
Number analyzed (Participants) | 9 | 10
participants | 6 | 8

3. Secondary Outcome: Proportion of Participants With an Infusion-related Reaction (IRR) on Day 168
Description: The proportion of patients having an infusion-related reaction as defined by Common Terminology Criteria (CTCAE), version 4 during or after receiving the first full 600mg dose infusion on week 168
Time Frame: during or after receiving the first full 600mg dose infusion on day 168.
Measure: Number; unit: participants
Arm/Group | Diphenhydramine | Cetirizine
Number analyzed (Participants) | 9 | 10
participants | 7 | 8

4. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) Score on Days 0, 14 and 168
Description: Patient reported outcome on Treatment Satisfaction Questionnaire for Medication. TSQM is administered within 2 hours after ocrelizumab (OCR) infusion, may be completed via phone to assess patient treatment satisfaction for the infusion. TSQM covers four domains: Global satisfaction, Effectiveness, Side effects, and Convenience. The scores are calculated for each of the subscales, ranging from 0 to 100. Higher score indicates higher satisfaction of the participant with the treatment and lower score indicates lower satisfaction of the participant with the treatment.
Time Frame: After the infusions on day 0, day 14, and day 168.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diphenhydramine | Cetirizine
Number analyzed (Participants) | 9 | 10
score on a scale
  Global Satisfaction- Day 0 | 88.0 (15.7) | 90.8 (9.99)
  Effectiveness- Day 0 | 78.7 (18.2) | 86.7 (11.2)
  Side Effects- Day 0 | 94.4 (11.0) | 100 (0)
  Convenience- Day 0 | 87.6 (13.9) | 96.1 (5.89)
  Global Satisfaction- Day 14 | 88.6 (14.7) | 93.3 (11.7)
  Effectiveness- Day 14 | 78.1 (14.0) | 91.9 (14.2)
  Side Effects- Day 14 | 92.7 (10.4) | 100 (0)
  Convenience- Day 14 | 90.3 (11.0) | 96.6 (7.33)
  Global Satisfaction- Day 168 | 91.7 (13.9) | 99.1 (2.67)
  Effectiveness- Day 168 | 87.5 (15.6) | 93.5 (10.0)
  Side Effects- day 168 | 95.8 (6.98) | 96.3 (11.0)
  Convenience- Day 168 | 94.4 (7.04) | 95.7 (10.9)

5. Secondary Outcome: Stanford Sleepiness Scale (SSS) Score on Days 0, 14, and 168
Description: Patient reported outcome on Stanford Sleepiness Score (SSS) administered prior to starting and within 2 hours after ocrelizumab (OCR) infusion, may be completed via phone. SSS measures sleepiness at specific times in a day. Participants will use a scale from 1 to 7 best representing their level of perceived sleepiness. The higher the score, the sleepier the subject and a lower score indicates the alertness of the subject.
Time Frame: after the infusions on day 0, day 14, and day 168.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diphenhydramine | Cetirizine
Number analyzed (Participants) | 9 | 10
score on a scale
  Day 0 | 3.11 (1.27) | 1.90 (0.876)
  Day 14 | 3.13 (1.13) | 2.00 (0.667)
  Day 168 | 2.50 (0.837) | 2.33 (1.00)

6. Secondary Outcome: Visual Analog Scale for Fatigue (VAS-F) Score on Days 0, 14 and 168
Description: Patient reported outcomes on Visual Analog Scale for Fatigue, administered prior to starting and within 2 hours after ocrelizumab (OCR) infusion, may be completed via phone. The scale consists of various items relating to the participants' experience of fatigue and energy. Fatigue subscale ranges from 0-10 and a higher the score represents a greater fatigue for the participant. Energy subscale ranges from 0-10 and a higher the score represents a greater energy as perceived by the participant.
Time Frame: after the infusions on day 0, day 14, and day 168.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diphenhydramine | Cetirizine
Number analyzed (Participants) | 9 | 10
score on a scale
  Fatigue- Day 0 | 4.10 (2.19) | 1.92 (2.13)
  Energy at Day 0 | 5.20 (1.35) | 6.28 (2.56)
  Fatigue- Day 14 | 3.95 (1.94) | 1.94 (1.12)
  Energy- Day 14 | 4.63 (1.98) | 6.08 (1.80)
  Fatigue- Day 168 | 3.52 (1.08) | 2.12 (2.12)
  Energy- Day 168 | 5.33 (2.66) | 5.82 (2.43)

7. Secondary Outcome: Modified Fatigue Impact Scale (MFIS) Score on Day 168
Description: Modified Fatigue Impact Scale (MFIS) administered after the 2nd dose of OCR. Subject answers 21 questions (9 physical, 10 cognitive, and 2 psychological items) related to fatigue in the past 4 weeks with choices of frequency: 0: Never, 1: Rarely, 2: Sometimes, 3: Often, or 4: Almost always. The total MFIS score ranges from 0 to 84. A higher total score represents greater fatigue as perceived by the participants.
Time Frame: at day 168.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diphenhydramine | Cetirizine
Number analyzed (Participants) | 8 | 10
score on a scale | 23.9 (15.9) | 18.3 (22.2)

8. Secondary Outcome: Multiple Sclerosis Impact Scale (MSIS-29) Score on Day168
Description: Multiple Sclerosis Impact Scale (MSIS-29) is administered after the 2nd dose of ocrelizumab (OCR) infusion to evaluate the physical and psychological impact of multiple sclerosis (MS). Participants rate their symptoms related to MS as 1-Not at all, 2-a little 3-Moderately or 4-Extremely on the two subscales, 20-item physical subscale and 9-item psychological subscale. The two subscales are scored by summing the responses across items, then converting to a 0-100 scale using a formula. For both subscales, higher scores indicate higher impact of MS or greater disability for the participant.
  Formula for physical impact subscale score: (100*(observed score-20))/ (100-20) Formula for psychological impact subscale score: (100*(observed score 9))/ (45-9)
Time Frame: at day 168.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diphenhydramine | Cetirizine
Number analyzed (Participants) | 8 | 10
score on a scale
  Physical Subscale | 19.7 (25.7) | 6.38 (9.31)
  Psychological Subscale | 13.0 (10.2) | 12.3 (14.1)

ADVERSE EVENTS:
Time Frame: The period during which all adverse events and serious adverse events collected began after the informed consent is obtained and ends 30 days following the last administration of study treatment or study discontinuation/termination, whichever is earlier, up to 28 weeks.
Arm/Group | Diphenhydramine | Cetirizine
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 7/9 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diphenhydramine (N=9) | Cetirizine (N=10)
Infusion-related reaction (Immune system disorders) | 5 | 6 — IRR after the first half of first dose 9300mg) of OCR infusion
Infusion-related reaction (Immune system disorders) | 6 | 8 — IRR after the first two infusions of dose 1 (each 300mg)
Infusion-related reaction (Immune system disorders) | 7 | 8 — Overall IRRs occurred at the end of the study after infusion of dose 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT04175834/Prot_SAP_000.pdf